CLINICAL TRIAL: NCT02120287
Title: Multicenter Phase II Study of Border Zone Stereotactic Radiosurgery With Bevacizumab in Patients With Recurrent or Progressive Glioblastoma Multiforme
Brief Title: Border Zone Stereotactic Radiosurgery With Bevacizumab in Patients With Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ajay Niranjan (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ajay Niranjan, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-063
Record Dates: First submitted 2014-01-10; First posted 2014-04-22 (Estimated); Results first posted 2019-04-25 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Glioblastoma Multiforme; Glioblastoma - Category
Keywords: Border Zone Stereotactic Radiosurgery; Bevacizumab; Recurrent Glioblastoma Multiforme; Progressive Glioblastoma Multiforme; Magnetic Resonance Spectroscopy; Glioblastoma; Brain Cancer; Brain Tumor; Radiosurgery
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Bevacizumab; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BZ-SRS with Bevacizumab (Experimental): All patients will receive Border Zone Stereotactic Radiosurgery (BZ-SRS) and additionally receive bevacizumab (10 mg/kg) one day before and then at day 14 followed by 10 mg/kg/day every 14 days until progression.
  One to 14 days before BZ- SRS procedure, patients at centers with MRS experience will undergo standard brain MRI /MRS
  Interventions: Drug: Bevacizumab; Procedure: Magnetic Resonance Spectroscopy (MRS); Procedure: Border Zone Stereotactic Radiosurgery (BZ-SRS)

INTERVENTIONS:
Drug: Bevacizumab — Patients will receive bevacizumab (10 mg/kg) one day before and then at day 14 followed by10 mg/kg/day every 14 days until progression.
  Other Names: Avastin
Procedure: Magnetic Resonance Spectroscopy (MRS) — Subjects will have MRS prior to BZ-SRS.
Procedure: Border Zone Stereotactic Radiosurgery (BZ-SRS) — The 'border zone' of the tumor will be targeted by SRS in a single session.
  Other Names: GammaKnife

SUMMARY:
This is a phase II study on the usage of stereotactic Gamma Knife radiosurgery as a boost to the tumor bed border zone in conjunction with the usage of bevacizumab.

DETAILED DESCRIPTION:
Glioblastoma Multiforme (GBM) is the most common primary brain tumor in adults. Unfortunately, despite aggressive surgery, radiation therapy (RT) and chemotherapy, the prognosis for this disease is poor. It is our hypothesis that GBM is a "local" disease wherein treatment failure is due to failure to eradicate tumor cells in the pathways along which the tumor eventually spreads (the "border zone").

The investigators hypothesize that treatment volume escalation will be successful at improving overall survival in patients with GBM when appropriate targeting and precision dose delivery is performed in a single treatment session. The 'border zone' of the tumor will be targeted for SRS (defined as a combination of the MRI volume of gadolinium enhancement plus up to 2 cm of the surrounding T2 volume). This represents the volume of tumor infiltrated white matter and is the route of GBM spread. Bevacizumab, a monoclonal antibody to vascular endothelial growth factor (VEGF), has been used with safety and clinical success with concomitant chemotherapy in solid tumors, including GBM.

The investigators further hypothesize that a combined approach of SRS with this VEGF inhibitor will be an effective strategy for GBM because bevacizumab will maximize the effects of radiation in the treated volume and potentially reduce radiation toxicity in the adjacent brain.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed glioblastoma multiforme, WHO grade IV astrocytoma.
2. Prior first-line treatment with surgery or biopsy followed by fractionated radiotherapy with concurrent temozolomide-containing chemotherapy is required for glioblastoma patients. Additional prior chemotherapy is allowed, without limitation on number of recurrences.
3. An interval of at least 2 months since completion of fractionated radiotherapy.
4. Age > 18 years
5. Life expectancy of at least 12 weeks.
6. Karnofsky Performance Status score (KPS) of ≥ 60
7. Documented recurrent disease; Disease must be evaluable, but does not need to be measurable; the target site for SRS does not need to be located in a previously-irradiated area.
8. All patients must have no restrictions to obtaining MRI with and without gadolinium contrast.
9. Adequate bone marrow, hepatic and renal function ; BUN < 25 and Cr < 1.7
10. Negative pregnancy test at the time of SRS in any patient who could be pregnant.
11. Willingness to forego additional therapy until evidence of disease progression

Exclusion Criteria:

1. General Medical Exclusions:

1. Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study.
2. Active malignancy, other than superficial basal cell and superficial squamous (skin) cell, or carcinoma in situ of the cervix within last 3 years.
3. Prior radiosurgery
4. Prior intracavitary irradiation or Gliadel wafers.

2. Disease-Specific Exclusions:

1. Inability to comply with protocol or study procedures
2. Prior treatment with bevacizumab.
3. Inability to undergo MRI with and without contrast administration.

3. Bevacizumab-Specific Exclusions:

1. Inadequately controlled hypertension.
2. Prior history of hypertensive crisis or hypertensive encephalopathy.
3. New York Heart Association (NYHA) Grade II or greater congestive heart failure.
4. History of myocardial infarction or unstable angina within 6 months prior to Day 1.
5. History of stroke or transient ischemic attack within 6 months prior to Day 1.
6. Significant vascular disease within 6 months prior to Day 1.
7. History of hemoptysis within 1 month prior to Day 1.
8. Evidence of bleeding diathesis or significant coagulopathy
9. Major surgical procedure, open biopsy, or significant traumatic injury within 14 days prior to Day 1 or anticipation of need for major non -cranial surgical procedure during the course of the study.
10. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1.
11. History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1.
12. Serious, non-healing wound, active ulcer, or untreated bone fracture.
13. Proteinuria
14. Known hypersensitivity to any component of bevacizumab
15. Pregnancy (positive pregnancy test) or lactation. Use of effective means of contraception (men and women) in subjects of child-bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-05; Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Niranjan, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- BZ-SRS With Bevacizumab: All patients received Border Zone Stereotactic Radiosurgery (BZ-SRS) and additionally received bevacizumab (10 mg/kg) one day before and then at day 14 followed by 10 mg/kg/day every 14 days until disease progression. One to 14 days before BZ- SRS procedure, patients at centers with MRS experience will undergo standard brain MRI /MRS. Patients will have MRS Magnetic Resonance Spectroscopy (MRS)prior to BZ-SRS. Border Zone Stereotactic Radiosurgery (BZ-SRS): The 'border zone' of the tumor will be targeted by SRS in a single session.
Period: Overall Study
Arm/Group | BZ-SRS With Bevacizumab
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with recurrent or Progressive Glioblastoma Multiforme who underwent treatment of border Zone Stereotactic Radiosurgery (BZ-SRS) with bevacizumab (10 mg/kg).
Arm/Group | BZ-SRS With Bevacizumab
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 62 [48.7 to 74.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: The number of months that a patient remains alive from the day first gamma knife surgery until the date of death or end of data collection for survival.
Time Frame: Up to 2 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BZ-SRS With Bevacizumab
Number analyzed (Participants) | 16
months | 11.73 [8.64 to 26.05]

2. Secondary Outcome: 6-month Progression-free Survival
Description: The proportion of patients who did not experience disease progression per RANO as of 6 months from the date of radiosurgery. RANO (Response Assessment in Neuro-Oncology) Response Criteria for Progression using imaging features: 25% or more increase in enhancing lesions despite stable or increasing steroid dose increase (significant) in non-enhancing FLAIR/T2W lesions, not attributable to other non-tumor causes any new lesions clinical features clinical deterioration (not attributable to other non-tumor causes and not due to steroid decrease). Proportion of patients for PFS = number of patients without disease at 6 months post radiosurgery / total number of patients.
Time Frame: At 6 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | BZ-SRS With Bevacizumab
Number analyzed (Participants) | 16
proportion of participants
  Death or disease progression ≤ 6mons of treatment | 0.438 [0.198 to 0.701]
  Alive or stable disease ≥ 6 months of treatment | 0.562 [0.299 to 0.802]

3. Secondary Outcome: 6-month Overall Survival
Description: The proportion of patients who remained alive as of 6 months from the date of radiosurgery. Proportion of patients for OS = number of patients alive at 6 months post radiosurgery / total number of patients.
Time Frame: At 6 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | BZ-SRS With Bevacizumab
Number analyzed (Participants) | 16
proportion of participants
  Death within 6 months of treatment | 0.0625 [0.0158 to 0.302]
  Alive after 6 months of treatment | 0.938 [0.698 to 0.998]

4. Secondary Outcome: CNS Toxicity
Description: The number of patients experiencing a CNS toxicity type occurring within 3 months of gamma knife surgery, as measured by RTOG/EORTC Acute Radiation Morbidity Scoring and the NCI CTCAE v4.0 for late toxicity.
Time Frame: Six months after SRS
Population: as for baseline characteristics
Measure: Number; unit: number of participants
Arm/Group | BZ-SRS With Bevacizumab
Number analyzed (Participants) | 16
number of participants
  Muscle Weakness Lower Limb | 1
  Fatigue and Dehydration | 1
  Spinal Fracture and Pain | 1

5. Secondary Outcome: Tumor Response
Description: Proportion of patients with a best response of CR, PR, SD, PD: number of patients with CR, PR, SD or PD / total number of patients evaluable for response to treatment of border zone Stereotactic Radiosurgery (BZ-SRS) with bevacizumab.
Time Frame: Up to 2 years
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | BZ-SRS With Bevacizumab
Number analyzed (Participants) | 16
Proportion of participants
  Complete Response | 0.077 [0.0019 to 0.360]
  Partial Response | 0.308 [0.091 to 0.614]
  Stable Disease | 0.538 [0.251 to 0.808]
  Progressed Disease | 0.077 [0.0019 to 0.360]

6. Secondary Outcome: Potential Value of Magnetic Resonance Spectroscopy (MRS)
Description: Improvement of border zone target selection and detection of therapeutic response of the derived treatment volumes between MRI and MRI+MRS (Magnetic Resonance Spectroscopy).
  This is presented as the number of patients for whom the derived treatment was changed as a result of the utilization of MRS.
Time Frame: Prior to radiosurgery
Population: Participants who received MRS (Magnetic Resonance Spectroscopy) scans prior to radiosurgery.
Measure: Number; unit: number of participants
Arm/Group | BZ-SRS With Bevacizumab
Number analyzed (Participants) | 11
number of participants | 0

7. Secondary Outcome: Karnofsky Performance Status
Description: The Karnofsky Performance Scale Index allows patients to be classified as to their functional impairment. This can be used to compare effectiveness of different therapies and to assess the prognosis in individual patients. Score range from 0 to 100; the lower the Karnofsky score, the worse the survival for most serious illnesses. A score of 100 would indicate 'Normal no complaints; no evidence of disease.' A score of 50 indicates 'Requires considerable assistance and frequent medical care.' A score of 0-10 would indicate 'Moribund; fatal processes progressing rapidly' and 'Death'.
Time Frame: At baseline (Week 0) prior to treatment administration
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | BZ-SRS With Bevacizumab
Number analyzed (Participants) | 16
participants
  Karnofsky Performance Status Score: 40 | 0
  Karnofsky Performance Status Score: 60 | 0
  Karnofsky Performance Status Score: 70 | 4
  Karnofsky Performance Status Score: 80 | 6
  Karnofsky Performance Status Score: 90 | 6
  Karnofsky Performance Status Score: 100 | 0

8. Secondary Outcome: Barthel's Index of Activities of Daily Living Assessment
Description: The Barthel Index consists items assessing the ability to achieve certain activities without assistance. It evaluates the ability of feeding, moving from wheelchair to bed and returning, doing personal toilet, getting on and off toilet,bathing self, walking on level surface, ascending and descending stairs, dressing, controlling bowels and controlling bladder. Scoring ranged from 0 (completely dependent) to 20 (completely independent) for this assessment. A maximal score of 20 indicating that a patient is fully independent in physical functioning, and a lowest score of 0 representing a totally dependent bed-ridden state.
Time Frame: At baseline (Week 0) prior to treatment administration
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BZ-SRS With Bevacizumab
Number analyzed (Participants) | 13
score on a scale | 17.77 [10.98 to 24.55]

9. Secondary Outcome: Barthel's Index of Activities of Daily Living Assessment
Description: as for outcome 8
Time Frame: At 8 weeks
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BZ-SRS With Bevacizumab
Number analyzed (Participants) | 10
score on a scale | 16.30 [5.16 to 27.44]

10. Secondary Outcome: Center for Epidemiological Studies Depression Scale (CES-D)
Description: An assessment comprised of 20 statements for which the participant is asked to indicate how often they have felt a certain way during the past week. SCORING: zero for answers of Rarely or none of the time (less than 1 day), 1 for answers of Some or a little of the time (1-2 days), 2 for answers of Occasionally or a moderate amount of time (3-4 days) the third column, 3 for answers of Most or all of the time (5-7 days). The scoring of positive items is reversed. Possible range of scores is zero to 60, with the higher scores indicating the presence of more depression symptomatology.
Time Frame: At baseline (Week 0) prior to treatment administration
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | BZ-SRS With Bevacizumab
Number analyzed (Participants) | 13
score on a scale | 17.0 [10.5 to 23.5]

11. Secondary Outcome: Center for Epidemiological Studies Depression Scale (CES-D)
Description: as for outcome 10
Time Frame: At 8 weeks
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | BZ-SRS With Bevacizumab
Number analyzed (Participants) | 9
score on a scale | 20.2 [12.2 to 28.3]

12. Secondary Outcome: Functional Assessment of Cancer - General (FACT-G)
Description: The FACT-G is a patient rated, 27-item compilation of general questions divided into 4 primary Quality of Life (QOL) sub-scales: physical well-being (PWB; 7-items, score range 0-28), social/family well-being (SWB; 7-items, score range 0-28), emotional well-being (EWB; 6-items, score range 0-24), and functional well-being (FWB; 7-items, score range 0-28). This tool represents the generic core questionnaire that are utilized in combination with cancer site-specific questionnaires, (FBrain, in this study) Overall score and four subscale scores with ranges and distributions that are sample-specific can be calculated.FACT-G is scored by summing the individual scale scores; higher scores indicate better quality of life. FACT-G uses 5-point rating scale ranging from (0) = Not at all; (1) = A little bit; (2) = Somewhat; (3) = Quite a bit; to (4) = Very much.The FACT-G total score is the sum of the four subscale scores (if least 80% completed) and has a possible range of 0-108 points.
Time Frame: At baseline (Week 0) prior to treatment administration
Population: Patients with recurrent or Progressive Glioblastoma Multiforme who underwent treatment of border Zone Stereotactic Radiosurgery (BZ-SRS) with bevacizumab (10 mg/kg). (NOTE: One participant did not complete the EWB section of the questionnaire. One participant did not complete the FWB section of the questionnaire.)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BZ-SRS With Bevacizumab
Number analyzed (Participants) | 14
score on a scale
  Physical Well-Being | 18.9 [14.9 to 22.8]
  Social Well-Being | 23.6 [22.0 to 25.3]
  Emotional Well-Being | 15.8 [12.4 to 19.3]
  Functional Well-Being | 16.8 [12.6 to 20.9]
  Total Well-Being | 75.8 [64.3 to 87.3]

13. Secondary Outcome: Functional Assessment of Cancer Therapy-General - General (FACT-G)
Description: as for outcome 12
Time Frame: At 8 weeks
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BZ-SRS With Bevacizumab
Number analyzed (Participants) | 10
score on a scale
  Physical Well-Being | 20.0 [17.3 to 22.7]
  Social Well-Being | 23.1 [20.9 to 25.3]
  Emotional Well-Being | 16.4 [12.9 to 19.9]
  Functional Well-Being | 15.8 [10.3 to 21.3]
  Total Well-Being | 75.3 [65.7 to 84.9]

14. Secondary Outcome: Functional Assessment of Cancer Therapy-Brain Specific Symptom Index (FACT-BrSI)
Description: The FACT-BrSI subscale, brain tumor specific version (2007), is a 15-item, patient completed, questionnaire.This brain subscale is used along with the core (general) questionnaire (FACT-G) that includes 27 items. Patients rate all items using a five-point Likert scale ranging from 0 "not at all" to 4 "very much." Overall, higher ratings suggest higher quality of life (QOL). The FACT BrSI has a range of 0-60, where a higher score indicates less symptomatology.
Time Frame: At baseline (Week 0) prior to treatment administration
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BZ-SRS With Bevacizumab
Number analyzed (Participants) | 14
score on a scale | 39.7 [32.5 to 47.0]

15. Secondary Outcome: Functional Assessment of Cancer Therapy-Brain Specific Symptom Index (FACT-BrSI)
Description: as for outcome 14
Time Frame: At 8 weeks
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BZ-SRS With Bevacizumab
Number analyzed (Participants) | 10
score on a scale | 40.5 [37.1 to 43.9]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | BZ-SRS With Bevacizumab
All-Cause Mortality (participants affected / at risk) | 14/16
Serious Adverse Events (participants affected / at risk) | 7/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BZ-SRS With Bevacizumab (N=16)
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Gait disturbance (General disorders) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cognitive disturbance (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 4
Confusion (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BZ-SRS With Bevacizumab (N=16)
Anemia (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Blurred vision (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 11
Gait disturbance (General disorders) | 2
General disorders and administration site conditions - Other, specify (General disorders) | 1
Pain (General disorders) | 5
Mucosal infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 3
Skin infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 3
Intraoperative musculoskeletal injury (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Cholesterol high (Investigations) | 2
Investigations - Other, specify (Investigations) | 2
Lymphocyte count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 4
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Cognitive disturbance (Nervous system disorders) | 4
Dysarthria (Nervous system disorders) | 2
Headache (Nervous system disorders) | 5
Nervous system disorders - Other, specify (Nervous system disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 2
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Personality change (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 5
Phlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT02120287/Prot_SAP_000.pdf